CLINICAL TRIAL: NCT06952374
Title: Mitral Valve Lithotripsy Using the SMARTWAVE Balloon for Severe Mitral Annular or Valvular Calcification (SMART-MAC): First in Human Study
Brief Title: Treating Severe Mitral Valve Annular or Valvular Calcification Using Shockwave Balloon SMARTWAVE
Acronym: SMARTMAC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Prince of Wales Hospital, Shatin, Hong Kong (Other)
Collaborators: Peijia Medical Technology (Suzhou) Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Dr So Chak Yu kent, Clinical assistant professor, Prince of Wales Hospital, Shatin, Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024.362
Record Dates: First submitted 2025-02-06; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Mitral Annulus Calcification; Rheumatic Heart Disease
Keywords: Mitral valve stenosis
MeSH Terms: conditions — Rheumatic Heart Disease; Mitral Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SmartWave (Experimental)
  Interventions: Device: SmartWave Lithotripsy balloon

INTERVENTIONS:
Device: SmartWave Lithotripsy balloon — ntravascular lithotripsy is an approved adjunct interventional therapy in treating calcified lesions to facilitate stenotic lesion opening in peripheral vascular disease and coronary artery disease. The off-label use of current peripheral lithotripsy balloon in mitral valve as a compassionate treatment or as an adjunct treatment before mitral balloon valvuloplasty and transcatheter mitral valve replacement has been reported with success . A possible mechanism is that lithotripsy preferentially impacts hard tissue, disrupts calcium, and leaves soft tissue undisturbed, improving valve pliability, preventing leaflet damage, and making subsequent valvuloplasty safer.

SUMMARY:
Mitral stenosis (MS) is a heavily symptomatic valvular heart disease. Common causes of MS included chronic rheumatic heart disease (CRHD) and mitral annular calcification (MAC). Current guideline recommends percutaneous balloon mitral valvuloplasty (PBMV) being the first line intervention for rheumatic MS with favorable anatomy. However, severely calcified mitral valve (i.e. those with Wilkins scores>8) makes the mitral valve non-pliable and carries high risk of severe mitral regurgitation (MR) (4-19%) with conventional balloon valvuloplasty. MAC is an increasingly recognized disease associated with atherosclerotic risk factors, and a well-recognized valve morphology that responses poorly with PBMV. Besides, conventional open-heart surgery for MAC-associated mitral valve dysfunction carries high mortality. Transcatheter mitral valve replacement with valve-in-MAC has become an alternative in treating these patients. However, valve-in-MAC is not always feasible and still carries operative and 30-day mortality.

Intravascular lithotripsy is an approved adjunct interventional therapy in treating calcified lesions to facilitate stenotic lesion opening in peripheral vascular disease and coronary artery disease. The off-label use of current peripheral lithotripsy balloon in mitral valve as a compassionate treatment or as an adjunct treatment before mitral balloon valvuloplasty and transcatheter mitral valve replacement has been reported with success . A possible mechanism is that lithotripsy preferentially impacts hard tissue, disrupts calcium, and leaves soft tissue undisturbed, improving valve pliability, preventing leaflet damage, and making subsequent valvuloplasty safer. However, the off-label use of multiple peripheral lithotripsy balloons in mitral valve is technically complicated.

SmartWave balloon was specifically designed lithotripsy balloon for calcified aortic stenosis. This first-in-human study aims to apply the SmartWave lithotripsy balloon in treating calcified mitral stenosis due to MAC or severely calcified rheumatic mitral valve.

DETAILED DESCRIPTION:
Mitral stenosis (MS) is a heavily symptomatic valvular heart disease. Common causes of MS included chronic rheumatic heart disease (CRHD) and mitral annular calcification (MAC). Current guideline recommends percutaneous balloon mitral valvuloplasty (PBMV) being the first line intervention for rheumatic MS with favorable anatomy. However, severely calcified mitral valve (i.e. those with Wilkins scores>8) makes the mitral valve non-pliable and carries high risk of severe mitral regurgitation (MR) (4-19%) with conventional balloon valvuloplasty. MAC is an increasingly recognized disease associated with atherosclerotic risk factors, and a well-recognized valve morphology that responses poorly with PBMV. Besides, conventional open-heart surgery for MAC-associated mitral valve dysfunction carries high mortality. Transcatheter mitral valve replacement with valve-in-MAC has become an alternative in treating these patients. However, valve-in-MAC is not always feasible and still carries operative and 30-day mortality.

Intravascular lithotripsy is an approved adjunct interventional therapy in treating calcified lesions to facilitate stenotic lesion opening in peripheral vascular disease and coronary artery disease. The off-label use of current peripheral lithotripsy balloon in mitral valve as a compassionate treatment or as an adjunct treatment before mitral balloon valvuloplasty and transcatheter mitral valve replacement has been reported with success . A possible mechanism is that lithotripsy preferentially impacts hard tissue, disrupts calcium, and leaves soft tissue undisturbed, improving valve pliability, preventing leaflet damage, and making subsequent valvuloplasty safer. However, the off-label use of multiple peripheral lithotripsy balloons in mitral valve is technically complicated.

SmartWave balloon was specifically designed lithotripsy balloon for calcified aortic stenosis. This first-in-human study aims to apply the SmartWave lithotripsy balloon in treating calcified mitral stenosis due to MAC or severely calcified rheumatic mitral valve.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 and
* Able to give procedure and study consent and
* Severe symptomatic mitral stenosis (MVA <1.5cm^2 derived by 3D planimetry or continuity equation or pressure half time) and
* Presence of mitral annular calcification or
* CRHD with severe leaflet calcification with Wilkins score >8

Exclusion Criteria:

* Baseline > moderate MR
* Intracardiac thrombus as visualized by TEE
* Pregnant patients. Female patients of childbearing potential must have a negative pregnancy test (per site standard test) within 7 days prior to index procedure.
* Active infection with bacteremia
* Current participation in another investigational drug or device study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-03-08 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Improvement in mitral valve area | Post-OP 6 and 12 month
  Immediate and sustained improvement in mitral valve area (MVA >1.5cm^2) without significant worsening of MR (> moderate)
Absence of peri-procedural complication | At and peri-procedure
  Absence of peri-procedural complication (death, stroke, myocardial infarction, cardiac tamponade, conversion to open heart) defined according to the Mitral Valve Academic Research Consortium

SECONDARY OUTCOMES:
Hemodynamic changes | Intra-operation
  Invasive haemodyanmic changes after each lithotripsy cycle
Mitral valve calcification level | Baseline and post-procedure up to 1 year
  Baseline and post-procedural mitral valve calcium distribution and volume determined by computed tomography
Symptom status change (New York Heart Aassociation functional class) | Baseline,Post-OP 1 month, 3 month, 6 month, 12 month
  Symptom status change assessed by New York Heart Aassociation functional class
Symptom status change (By Kansas City Cardiomyopathy Questionnaire-12) | Baseline,Post-OP 1 month, 3 month, 6 month, 12 month
  Symptom status change assessed by Kansas City Cardiomyopathy Questionnaire-12
Debris histology | peri-operation
  Sentinel captured debris will be collected and sent for histology analysis to look for signs of tissue damage or calcification break off.
NTproBNP | baseline, post-operation, Post-OP 1, 3, 6, 12 month
  Change of NTproBNP
Lung Fluid | baseline, Post-OP 1, 3, 6, 12 month
  Change in lung fluid percentage
Major Adverse Cardiac Event | 6 month and 12 month post-operation
  6 month and 12 month clinical event (death, heart failure hospitalization, stroke, myocardial infarction, mitral valve reintervention)

CONTACTS AND LOCATIONS:
Overall Officials: Kent So, MbChB, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Shatin, New Territories, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Stone GW, Adams DH, Abraham WT, Kappetein AP, Genereux P, Vranckx P, Mehran R, Kuck KH, Leon MB, Piazza N, Head SJ, Filippatos G, Vahanian AS; Mitral Valve Academic Research Consortium (MVARC). Clinical Trial Design Principles and Endpoint Definitions for Transcatheter Mitral Valve Repair and Replacement: Part 2: Endpoint Definitions: A Consensus Document From the Mitral Valve Academic Research Consortium. J Am Coll Cardiol. 2015 Jul 21;66(3):308-321. doi: 10.1016/j.jacc.2015.05.049. PMID 26184623
- [Background] Giustino G, Fang JX, Villablanca PA, Wang DD, Sturla N, Lee JC, O'Neill BP, Frisoli T, O'Neill WW, Engel-Gonzalez P. Intravascular Lithotripsy-Facilitated Balloon Valvuloplasty for Severely Calcified Mitral Valve Stenosis. JACC Cardiovasc Interv. 2024 Jan 22;17(2):326-327. doi: 10.1016/j.jcin.2023.10.015. Epub 2023 Dec 20. No abstract available. PMID 38127026
- [Background] Sharma A, Kelly R, Mbai M, Chandrashekhar Y, Bertog S. Transcatheter Mitral Valve Lithotripsy as a Pretreatment to Percutaneous Balloon Mitral Valvuloplasty for Heavily Calcified Rheumatic Mitral Stenosis. Circ Cardiovasc Interv. 2020 Jul;13(7):e009357. doi: 10.1161/CIRCINTERVENTIONS.120.009357. Epub 2020 Jul 17. No abstract available. PMID 32674681
- [Background] Eng MH, Villablanca P, Wang DD, Frisoli T, Lee J, O'Neill WW. Lithotripsy-Facilitated Mitral Balloon Valvuloplasty for Senile Degenerative Mitral Valve Stenosis. JACC Cardiovasc Interv. 2019 Aug 12;12(15):e133-e134. doi: 10.1016/j.jcin.2019.05.026. Epub 2019 Jul 17. No abstract available. PMID 31326427
- [Background] Tepe G, Brodmann M, Werner M, Bachinsky W, Holden A, Zeller T, Mangalmurti S, Nolte-Ernsting C, Bertolet B, Scheinert D, Gray WA; Disrupt PAD III Investigators. Intravascular Lithotripsy for Peripheral Artery Calcification: 30-Day Outcomes From the Randomized Disrupt PAD III Trial. JACC Cardiovasc Interv. 2021 Jun 28;14(12):1352-1361. doi: 10.1016/j.jcin.2021.04.010. PMID 34167675
- [Background] Rodriguez-Leor O, Cid-Alvarez AB, Lopez-Benito M, Gonzalo N, Vilalta V, Diarte de Miguel JA, Lopez LF, Jurado-Roman A, Diego A, Oteo JF, Cuellas C, Trillo R, Travieso A, Alfonso F, Carrillo X, Vegas-Valle JM, Cortes-Villar C, Pascual I, Munoz Camacho JF, Flores X, Vera-Vera S, Moreu J, Barreira de Sousa G, Marti D, Jimenez-Mazuecos J, Fuertes M, Ocaranza R, de la Torre Hernandez JM, Lozano F, Solana Martinez SG, Gomez-Lara J, Perez de Prado A; REPLICA-EPIC18 Investigators. A Prospective, Multicenter, Real-World Registry of Coronary Lithotripsy in Calcified Coronary Arteries: The REPLICA-EPIC18 Study. JACC Cardiovasc Interv. 2024 Mar 25;17(6):756-767. doi: 10.1016/j.jcin.2023.12.018. Epub 2024 Feb 21. PMID 38385926
- [Background] Kereiakes DJ, Hill JM, Shlofmitz RA, Klein AJ, Riley RF, Price MJ, Herrmann HC, Bachinsky W, Waksman R, Stone GW; Disrupt CAD III Investigators. Intravascular Lithotripsy for Treatment of Severely Calcified Coronary Arteries: 2-Year Results-Disrupt CAD III Study. JACC Cardiovasc Interv. 2023 Oct 9;16(19):2472-2474. doi: 10.1016/j.jcin.2023.07.010. Epub 2023 Sep 6. No abstract available. PMID 37676225
- [Background] Ali ZA, Kereiakes D, Hill J, Saito S, Di Mario C, Honton B, Gonzalo N, Riley R, Maehara A, Matsumura M, Stone GW, Shlofmitz R. Safety and Effectiveness of Coronary Intravascular Lithotripsy for Treatment of Calcified Nodules. JACC Cardiovasc Interv. 2023 May 8;16(9):1122-1124. doi: 10.1016/j.jcin.2023.02.015. Epub 2023 Apr 5. No abstract available. PMID 37029020
- [Background] Maisano F, Taramasso M. Mitral valve-in-valve, valve-in-ring, and valve-in-MAC: the Good, the Bad, and the Ugly. Eur Heart J. 2019 Feb 1;40(5):452-455. doi: 10.1093/eurheartj/ehy725. No abstract available. PMID 30476035
- [Background] Guerrero ME, Eleid MF, Wang DD, Pursnani A, Kodali SK, George I, Palacios I, Russell H, Makkar RR, Kar S, Satler LF, Rajagopal V, Dangas G, Tang GHL, McCabe JM, Whisenant BK, Fang K, Balan P, Smalling R, Kaptzan T, Lewis B, Douglas PS, Hahn RT, Thaden J, Oh JK, Leon M, O'Neill W, Rihal C. 5-Year Prospective Evaluation of Mitral Valve-in-Valve, Valve-in-Ring, and Valve-in-MAC Outcomes: MITRAL Trial Final Results. JACC Cardiovasc Interv. 2023 Sep 25;16(18):2211-2227. doi: 10.1016/j.jcin.2023.06.041. PMID 37758379
- [Background] Guerrero M, Wang DD, Pursnani A, Eleid M, Khalique O, Urena M, Salinger M, Kodali S, Kaptzan T, Lewis B, Kato N, Cajigas HM, Wendler O, Holzhey D, Pershad A, Witzke C, Alnasser S, Tang GHL, Grubb K, Reisman M, Blanke P, Leipsic J, Williamson E, Pellikka PA, Pislaru S, Crestanello J, Himbert D, Vahanian A, Webb J, Hahn RT, Leon M, George I, Bapat V, O'Neill W, Rihal C. A Cardiac Computed Tomography-Based Score to Categorize Mitral Annular Calcification Severity and Predict Valve Embolization. JACC Cardiovasc Imaging. 2020 Sep;13(9):1945-1957. doi: 10.1016/j.jcmg.2020.03.013. Epub 2020 May 13. PMID 32417332
- [Background] Chehab O, Roberts-Thomson R, Bivona A, Gill H, Patterson T, Pursnani A, Grigoryan K, Vargas B, Bokhary U, Blauth C, Lucchese G, Bapat V, Guerrero M, Redwood S, Prendergast B, Rajani R. Management of Patients With Severe Mitral Annular Calcification: JACC State-of-the-Art Review. J Am Coll Cardiol. 2022 Aug 16;80(7):722-738. doi: 10.1016/j.jacc.2022.06.009. PMID 35953138
- [Background] Wilkins GT, Weyman AE, Abascal VM, Block PC, Palacios IF. Percutaneous balloon dilatation of the mitral valve: an analysis of echocardiographic variables related to outcome and the mechanism of dilatation. Br Heart J. 1988 Oct;60(4):299-308. doi: 10.1136/hrt.60.4.299. PMID 3190958
- [Background] Iung B, Nicoud-Houel A, Fondard O, Hafid Akoudad, Haghighat T, Brochet E, Garbarz E, Cormier B, Baron G, Luxereau P, Vahanian A. Temporal trends in percutaneous mitral commissurotomy over a 15-year period. Eur Heart J. 2004 Apr;25(8):701-7. doi: 10.1016/j.ehj.2004.02.026. PMID 15084376
- [Background] Writing Committee Members; Otto CM, Nishimura RA, Bonow RO, Carabello BA, Erwin JP 3rd, Gentile F, Jneid H, Krieger EV, Mack M, McLeod C, O'Gara PT, Rigolin VH, Sundt TM 3rd, Thompson A, Toly C. 2020 ACC/AHA Guideline for the Management of Patients With Valvular Heart Disease: A Report of the American College of Cardiology/American Heart Association Joint Committee on Clinical Practice Guidelines. J Am Coll Cardiol. 2021 Feb 2;77(4):e25-e197. doi: 10.1016/j.jacc.2020.11.018. Epub 2020 Dec 17. No abstract available. PMID 33342586